CLINICAL TRIAL: NCT00436917
Title: Zoledronic Acid for Treatment of Osteopenia and Osteoporosis in Women With Primary Breast Cancer Undergoing Adjuvant Aromatase Inhibitor (Letrozole) Therapy
Brief Title: Zoledronate in Treating Osteopenia or Osteoporosis in Postmenopausal Women Receiving Letrozole for Stage I, Stage II, or Stage IIIA Primary Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC05C8; P30CA015083 (NIH); MC05C8 (Other: Mayo Clinic Cancer Center); 2330-05 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2016-04

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; osteoporosis
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Zoledronic Acid; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- zoledronic acid (Experimental): 4 mg 15 minutes IV infusion. If creatinine clearance is ≤ 60, dosage should be adjusted as follows:CrCl 50-60: 3.5 mg; CrCl 40-49: 3.3 mg; CrCl 30-39: 3.0 mg.
  Interventions: Drug: zoledronic acid; Procedure: Letrozole as adjuvant therapy

INTERVENTIONS:
Drug: zoledronic acid — zoledronic acid
  Other Names: Zometa®
Procedure: Letrozole as adjuvant therapy — standard care
  Other Names: Femara®

SUMMARY:
RATIONALE: Zoledronate may reduce bone loss in patients receiving letrozole for breast cancer.

PURPOSE: This clinical trial is studying how well zoledronate works in treating osteopenia or osteoporosis in postmenopausal women receiving letrozole for stage I, stage II, or stage IIIA primary breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess changes in total lumbar spine bone mineral density (BMD) from baseline to 12 months in postmenopausal women treated with zoledronate for osteopenia or osteoporosis and letrozole for hormone receptor-positive, stage I-IIIA primary breast cancer.

Secondary

* Determine changes in total lumbar spine BMD from baseline to 2, 3, 4, and 5 years in these patients.
* Determine changes in femoral neck BMD from baseline to 1, 2, 3, 4, and 5 years in these patients.
* Determine time to disease progression in these patients.

OUTLINE: This is an open-label, multicenter study.

* Adjuvant aromatase inhibitor therapy: Patients receive oral letrozole daily for up to 5 years in the absence of disease progression or unacceptable toxicity.
* Osteoporosis management: Patients receive zoledronate IV over 15 minutes on day 1. Patients also receive oral elemental calcium twice daily and oral vitamin D daily for 6 months. Treatment repeats every 6 months for up to 5 years in the absence of disease progression or unacceptable toxicity.

Patients undergo total lumbar spine and hip (femoral neck) bone density testing by dual energy x-ray absorptiometry (DXA) at baseline and annually for 5 years.

After completion of study therapy, patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized breast cancer

  * Stage I-IIIA disease
  * Adequately treated breast cancer

    * No clinical or radiological evidence of recurrent or metastatic disease
* Baseline total lumbar spine or femoral neck bone mineral density T-score < -2.0 standard deviation (e.g., a patient with a T score of -2.1 is eligible)
* Hormone-receptor status:

  * Estrogen receptor and/or progesterone receptor-positive breast cancer

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal, defined by 1 of the following criteria:

  * Age > 55 years with cessation of menses
  * Age ≤ 55 years with spontaneous cessation of menses for > 1 year
  * Age ≤ 55 years with spontaneous cessation of menses for ≤ 1 year, but amenorrheic (e.g., spontaneous or secondary to hysterectomy), AND has postmenopausal estradiol levels
  * Bilateral oophorectomy
* ECOG performance status 0-2
* Life expectancy ≥ 5 years
* WBC ≥ 3,000/mm³ OR granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Creatinine < 2.0 mg/dL
* Creatinine clearance ≥ 45 mL/min
* No hypercalcemia (i.e., calcium level > 1 mg/dL above ULN) OR hypocalcemia (i.e., calcium level > 0.5 mg/dL below lower limit of normal) within the past 6 months
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other nonmalignant systemic diseases, including any of the following:

  * Uncontrolled infection
  * Uncontrolled diabetes mellitus
  * Uncontrolled thyroid dysfunction
  * Disease affecting bone metabolism (hyperparathyroidism, hypercortisolism, Paget's disease, osteogenesis imperfecta)
  * Malabsorption syndrome
* No uncontrolled seizure disorders associated with falls
* No known hypersensitivity to zoledronate or other bisphosphonates, letrozole, calcium, or vitamin D
* No concurrent active dental problems, including any of the following:

  * Infection of the teeth or jawbone (maxillary or mandibular)
  * Dental or fixture trauma
  * Prior or current diagnosis of osteonecrosis of the jaw
  * Exposed bone in the mouth
  * Slow healing after dental procedures
* No contraindication to spine dual energy x-ray absorptiometry (DXA) as defined by any of the following:

  * History of surgery at the lumbosacral spine, with or without implantable devices
  * Scoliosis with a Cobb angle > 15 degrees at the lumbar spine
  * Immobility, hyperostosis, or sclerotic changes at the lumbar spine, or evidence of sclerotic abdominal aorta sufficient to interfere with DXA scan
  * Disease of the spine that would preclude the proper acquisition of a lumbar spine DXA
* No condition that would preclude study follow-up or compliance
* No psychiatric illness that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

* More than 3 weeks since prior and no other concurrent oral bisphosphonates
* No prior intravenous bisphosphonates
* No prior aromatase inhibitor therapy
* More than 6 months since prior anabolic steroids or growth hormone
* More than 2 weeks since prior and no concurrent inhibitor of osteoclastic bone resorption (e.g., calcitonin, mithramycin, or gallium nitrate)
* More than 30 days since prior systemic investigational drug and/or device
* More than 7 days since prior topical investigational drug
* More than 6 weeks since prior and no concurrent dental or jaw surgery (e.g., extraction, implants)
* Concurrent short-term corticosteroid therapy allowed
* No concurrent sodium fluoride, parathyroid hormone, or tibolone
* No other concurrent investigational drug or device

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2016-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Hines, MD, Study Chair — Mayo Clinic; Charles L. Loprinzi, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Result] Hines SL, Sloan JA, Atherton PJ, Perez EA, Dakhil SR, Johnson DB, Reddy PS, Dalton RJ, Mattar BI, Loprinzi CL. Zoledronic acid for treatment of osteopenia and osteoporosis in women with primary breast cancer undergoing adjuvant aromatase inhibitor therapy. Breast. 2010 Apr;19(2):92-6. doi: 10.1016/j.breast.2009.12.001. Epub 2010 Jan 15. PMID 20079640

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty participants were recruited between June 2006 and July 2007 at 6 individual sites participating in the Mayo Clinic Cancer Research Consortium (MCCRC).
Groups:
- Zoledronic Acid: 4 mg intravenously over 15 minutes every 6 months (until disease progression or for 5 years)
Period: Overall Study
Arm/Group | Zoledronic Acid
Started | 53 (7 participants (1 cancellation, 1 major violation, 5 ineligibles) were excluded from all analysis.)
Completed | 32
Not Completed | 21
Not completed — Withdrawal by Subject | 13
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Treatment for polymyalgia rheumatic | 1
Not completed — Increased creatinine | 1
Not completed — Personal conflicts of patient | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0
Prior tamoxifen [Number; unit: participants]
  Yes | 24
  No | 29
Duration of tamoxifen use [Number; unit: participants]
  Missing | 29
  <=2 years | 4
  >2 years | 20
Time since tamoxifen ended [Number; unit: participants]
  Missing | 29
  <1 year | 20
  >=1 year | 4
Prior chemotherapy [Number; unit: participants]
  Yes | 20
  No | 33
Previous fracture by history or X-ray [Number; unit: participants]
  Yes | 7
  No | 46
Bone Mineral Density Measurement in Lumbar Spine [Mean (Standard Deviation); unit: g/cm2] — Baseline bone mineral density measurement in lumbar spine for the 30 participants analyzed in primary analysis.
  g/cm2 | 0.86 (0.12)

OUTCOME MEASURES:

1. Primary Outcome: Average Intra-patient Change in Total Lumbar Spine (L1 to L4) Bone Mineral Density (BMD)
Description: Change: BMD values at twelve months post study entry minus BMD values at baseline, expressed as a percentage of the baseline value.
Time Frame: Baseline and 1 year
Population: The primary analysis is performed on data where participants had the same baseline and 1 year BMD Lumbar Spine measurement location (L1-L4, L2-L4 or 'other Lumbar Spine')
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 30
Percentage of the baseline value | 2.66 [1.27 to 4.62]
Statistical Analysis 1: Comparison: Zoledronic Acid; A sample of 60 participants was estimated to provide percentage statistics accuracy to within 13% with 95% confidence; Test type: Superiority or Other; p = 0.01, Kruskal-Wallis

2. Secondary Outcome: Average Intra-patient Change in Total Lumbar Spine (L1 to L4) Bone Mineral Density (BMD) at Year 2 Post Study Entry
Description: Change: BMD values at year 2 post study entry minus BMD values at baseline, expressed as a percentage of the baseline value.
Time Frame: Baseline and 2 year
Population: Analysis was performed on data where participants had the same baseline and 2 year BMD Lumbar Spine measurement location (L1-L4, L2-L4 or 'other Lumbar Spine')
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 27
Percentage of the baseline value | 4.94 [2.20 to 7.68]

3. Secondary Outcome: Average Intra-patient Change in Total Lumbar Spine (L1 to L4) Bone Mineral Density (BMD) at Year 3 Post Study Entry
Description: Change: BMD values at year 3 post study entry minus BMD values at baseline, expressed as a percentage of the baseline value.
Time Frame: Baseline and 3 year
Population: Analysis was performed on data where participants had the same baseline and 3 year BMD Lumbar Spine measurement location (L1-L4, L2-L4 or 'other Lumbar Spine')
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 22
Percentage of the baseline value | 6.20 [3.74 to 8.66]

4. Secondary Outcome: Average Intra-patient Change in Total Lumbar Spine (L1 to L4) Bone Mineral Density (BMD) at Year 4 Post Study Entry
Description: Change: BMD values at year 4 post study entry minus BMD values at baseline, expressed as a percentage of the baseline value.
Time Frame: Baseline and 4 year
Population: Analysis was performed on data where participants had the same baseline and 4 year BMD Lumbar Spine measurement location (L1-L4, L2-L4 or 'other Lumbar Spine')
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 13
Percentage of the baseline value | 6.99 [0.80 to 13.18]

5. Secondary Outcome: Average Intra-patient Change in Total Lumbar Spine (L1 to L4) Bone Mineral Density (BMD) at Year 5 Post Study Entry
Description: Change: BMD values at year 5 post study entry minus BMD values at baseline, expressed as a percentage of the baseline value.
Time Frame: Baseline and 5 year
Population: Analysis was performed on data where participants had the same baseline and 5 year BMD Lumbar Spine measurement location (L1-L4, L2-L4 or 'other Lumbar Spine')
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 11
Percentage of the baseline value | 11.71 [2.43 to 21.0]

6. Secondary Outcome: Average Intra-patient Change in Femoral Neck Bone Mineral Density (BMD) at Year 1 Post Study Entry
Description: Change: BMD values at year 1 post study entry minus BMD values at baseline, expressed as a percentage of the baseline value.
Time Frame: Baseline and 1 year
Population: Analysis was performed on data where participants had the same baseline and 1 year BMD Femoral Neck measurement location (Left femoral, right femoral)
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 32
Percentage of the baseline value | 5.66 [1.30 to 10.02]

7. Secondary Outcome: Average Intra-patient Change in Femoral Neck Bone Mineral Density (BMD) at Year 2 Post Study Entry
Description: as for outcome 2
Time Frame: Baseline and 2 year
Population: Analysis was performed on data where participants had the same baseline and 2 year BMD Femoral Neck measurement location (Left femoral, right femoral)
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 29
Percentage of the baseline value | 10.47 [2.14 to 18.80]

8. Secondary Outcome: Average Intra-patient Change in Femoral Neck Bone Mineral Density (BMD) at Year 3 Post Study Entry
Description: as for outcome 3
Time Frame: Baseline and 3 year
Population: Analysis was performed on data where participants had the same baseline and 3 year BMD Femoral Neck measurement location (Left femoral, right femoral)
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 28
Percentage of the baseline value | 8.44 [3.45 to 13.44]

9. Secondary Outcome: Average Intra-patient Change in Femoral Neck Bone Mineral Density (BMD) at Year 4 Post Study Entry
Description: as for outcome 4
Time Frame: Baseline and 4 year
Population: Analysis was performed on data where participants had the same baseline and 4 year BMD Femoral Neck measurement location (Left femoral, right femoral)
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 14
Percentage of the baseline value | 4.49 [-0.98 to 9.96]

10. Secondary Outcome: Average Intra-patient Change in Femoral Neck Bone Mineral Density (BMD) at Year 5 Post Study Entry
Description: as for outcome 5
Time Frame: Baseline and 5 year
Population: Analysis was performed on data where participants had the same baseline and 5 year BMD Femoral Neck measurement location (Left femoral, right femoral)
Measure: Mean (95% Confidence Interval); unit: Percentage of the baseline value
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 14
Percentage of the baseline value | 4.54 [-3.18 to 12.26]

11. Secondary Outcome: Maximum-Grade Toxicity Incidence at Least Possibly Related to Study Medications
Description: Adverse events were assessed per NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. Grade 1=Mild, Grade 2=Moderate.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 53
Participants
  Grade 1 Arthralgia | 7
  Grade 2 Arthralgia | 4
  Grade 3 Arthralgia | 1
  Grade 1 Creatinine Increase | 7
  Grade 2 Creatinite increase | 2
  Grade 2 Desquamating Rash | 1
  Grade 2 Headache | 1
  Grade 2 Hot flashes | 3
  Grade 1 Nausea | 2
  Grade 3 Pain in extremity | 1
  Grade 1 Fever | 2
  Grade 1 Vomiting | 1
  Grade 1 Musculoskeletal disorder | 1
  Grade 2 Urogenital disorder | 1

12. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from date of randomization to the documentation of disease progression.
Time Frame: Up to 5 years
Population: None of the participants had disease progression.
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected every 6 months on treatment up to 5 years.
Description: One participant was excluded from adverse event reporting due to the adverse event data was not available beyond the baseline time point. Adverse event data were collected every 6 months on treatment up to 5 years.
Arm/Group | Zoledronic Acid
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 1/52
Other Adverse Events (participants affected / at risk) | 45/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=52)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=52)
Nausea (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Creatinine increased (Investigations) | 11 (31)
INR increased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 (128)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No